CLINICAL TRIAL: NCT03175536
Title: Comparing Patient-Centered Outcomes for Adults and Children With Asthma in High-Deductible Health Plans With and Without Preventive Drug Lists
Brief Title: Asthma in Families Facing Out-of-pocket Requirements With Deductibles
Acronym: AFFORD
Status: Completed | Type: Observational
Sponsor: Harvard Pilgrim Health Care (Other)
Collaborators: Harvard School of Public Health (HSPH) (Other); Asthma and Allergy Foundation of America (Other); Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: PCORI-IHS-1602-34331; IHS-1602-34331 (Other Grant/Funding Number: PCORI)
Record Dates: First submitted 2017-05-23; First posted 2017-06-05 (Actual); Results first posted 2024-09-03 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-04

CONDITIONS: Asthma
Keywords: high-deductible health plan; medication adherence; out-of-pocket costs; preventive drug list; value-based insurance design
MeSH Terms: conditions — Asthma; Medication Adherence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- HDHP with PDL: Enrollees switched from a health savings account (HSA)-eligible high-deductible health plan (HDHP) without a preventive drug list (PDL) to a HSA-HDHP with a PDL
  Interventions: Other: HDHP with PDL
- HDHP without PDL: Enrollees who stayed in a HSA-HDHP without a PDL.
- traditional plan: Enrollees who remained in a traditional health plan with a deductible < $500

INTERVENTIONS:
Other: HDHP with PDL — Enrollment in a Health Savings Account-eligible high-deductible health plan with an annual individual deductible of >$1000 that includes a preventive drug list (a list of certain chronic medications that are exempt from the deductible)
  Groups: HDHP with PDL

SUMMARY:
Asthma is one of the most common chronic diseases in the U.S. Despite guidelines, adherence to recommended controller medications is low. Cost is an important barrier to adherence. Employers are increasingly adopting high-deductible health plans (HDHPs) which require deductibles of > $1,000 per individual/$2,000 per family each year. In HDHPs with Health Savings Accounts (HSAs), most medications and non-preventive care must be paid out-of-pocket (OOP) until the deductible is reached. The lower premiums of HSA-HDHPs are appealing, but the high level of OOP costs can lead patients to forgo needed care. HSA-HDHPs can exempt preventive care from the deductible, and employers can add Preventive Drug Lists (PDLs) which exempt certain chronic medications from the deductible (including asthma medications), making them free. PDLs have the potential to improve controller medication use, which could prevent negative health outcomes and reduce cost-related trade-offs for families.

The goal of this research is to evaluate the impact of these two developments in the health insurance market -- HSA-HDHPs and PDLs -- on medication use and clinical outcomes for adults and children with asthma. To do this, tteh investigators will first conduct in-depth interviews with patients with asthma and parents of children with asthma who have HDHPs and traditional plans. Interviews will collect patient-reported data on how patients and their families navigate their insurance plan and make health care decisions when faced with OOP costs. Findings from the interviews will inform analyses of data from a large national health plan from 2004-2017. Investigators will select adults and children with asthma whose employer switched them from traditional plans or HSA-HDHPs without PDLs to HSA-HDHPs with or without a PDL. Analyses will examine changes in asthma medication use, emergency department (ED) visits, hospitalizations, and OOP costs before and after changing plans compared to similar patients who did not switch to a HSA-HDHP. The study aims to: 1) understand health care decision making and experiences of families with asthma with HDHPs; 2) examine the impact of HSA-HDHPs with and without PDLs on use of asthma medications and asthma-related ED visits and hospitalizations; 3) examine the extent to which the response to HSA-HDHPs and PDLs is affected by the presence of other family members with asthma or other chronic conditions; 4) examine the impact of HSA-HDHPs with and without PDLs on OOP costs for families.

DETAILED DESCRIPTION:
Background and Significance Asthma is one of the most common serious chronic diseases of adults and children in the United States. Despite guidelines and evidence, adherence to recommended asthma controller medications is low. Cost is an important barrier to non-adherence to asthma medications. Employers are increasingly adopting high-deductible health plans (HDHPs) particularly those that qualify for Health Savings Accounts (HSAs), which subject most medications to deductibles rather than copayments as in traditional coverage. HSA-HDHPs can thus lead to forgone care due to cost, including clinically appropriate services such as asthma medications. As a response, value-based insurance designs (VBID) have been proposed to promote high-value care by reducing or eliminating cost-sharing for these services. One common example is a Preventive Drug List (PDL) that can accompany HSA-HDHPs, which exempts certain chronic medications from the deductible to promote adherence. Many PDLs include asthma controller and rescue medications. With the increasing prevalence of HSA-HDHPs, PDLs have the potential to improve controller medication adherence for both adults and children.

Study Aims: The goal of this research is to provide needed evidence on the impact of two important developments in the health insurance landscape, HSA-HDHPs and PDLs, and whether PDLs can mitigate cost barriers associated with HSA-HDHPs and improve patient-centered outcomes for adults and children with asthma. The Aims of this research are:

1. To understand health care decision making and experiences of families with asthma with HSA-HDHPs and PDLs.
2. To examine the impact of HSA-HDHPs with and without PDLs on use of asthma controller and rescue medications, and on adverse clinical outcomes (asthma-related ED visits and hospitalizations), overall and for vulnerable subgroups (low-income and racial/ethnic minority patients).
3. To examine the extent to which the response to HSA-HDHPs and PDLs is affected by the presence of other family members with asthma or other chronic conditions.
4. To examine the impact of HSA-HDHPs with and without PDLs on OOP costs for patients and families with asthma.

Sources of Data

Aim 1. This study will collect patient-reported data through in-depth qualitative phone interviews

Aims 2-4 will use 14 years (2004-2017) of enrollment and claims data from a large U.S. commercial health plan

Study Population

The Aim 1 study population will consist of adults with asthma and parents of children with asthma. Eligible participants will be those who are currently enrolled in employer-sponsored health insurance plans (high-deductible plans with and without a PDL, or traditional plans).

The health plan population will be identified through enrollment and claims data from Harvard Pilgrim Health Care (HPHC). Eligible patients will include adults aged 18-64 and children aged 4-17 years with a diagnosis of asthma. Patients will be selected if they have been enrolled in an employer-sponsored HSA-HDHP with or without a PDL, or a traditional plan without a high deductible, for the prior year. Among those eligible in each sub-group, the investigators will randomly select 9 from each cell to send a recruitment mailing, for a total of 81 patients or parents invited to participate.

A population from the Asthma and Allergy Foundation of America (AAFA) will be recruited through postings to AAFA's Asthma Online Community, Educational Support Group, email list serve, Facebook page, and newsletters.

For Aims 2-4, the study population will consist of adults aged 18-64 years and children aged 4-17 years with asthma. Study subjects must have spent a year in a traditional health plan with no or low deductibles prior to the switch to an HSA-HDHP without a PDL, or in a HSA-HDHP without a PDL prior to switching to an HSA-HDHP with PDL, and then remain enrolled for at least one year post-switch. Control group members spend a year in a traditional plan or HDHP without PDL then remain in that plan for at least another 12 months.

Enrollees over age 64 who are eligible for Medicare will be excluded. The investigators will identify members with asthma during the baseline year using the same claims-based algorithm in which an asthma diagnosis will be defined as having at least one inpatient or two outpatient claims in the prior year with a diagnosis of asthma based on International Classification of Diseases (ICD) 9 and 10 codes for asthma.

Eligible employers are those that offer only one plan type in a given benefit year: 1) traditional Health Maintenance Organization/Preferred Provider Organization/Point of Service plans (deductibles <$1000, copayments of <$50 for most services, tiered copayments for medicines); 2) HSA-HDHPs without PDLs; or 3) HSA-HDHPs with PDLs. The investigators will select "full-replacement" employers that replace a traditional plan or HSA-HDHP without PDL with an HSA-HDHP without PDL or HSA-HDHP with PDL, respectively, for all employees at a given point in time; matched comparison employers will include those that keep all employees in their prior plan.

Outcomes

Aim 1 qualitative interviews will assess patient and family experiences across a number of domains related to asthma health care decision making and outcomes in HDHPs.

The primary study outcomes for Aims 2-4 are the claims-based measures of asthma medication use, outcomes, and OOP costs listed below, measured at the individual level. See section on primary outcomes for details,

Predictors and Covariates

The primary predictor variables include study period and insurance type. Study period indicates the one-year period before or up to three years after the index date. Insurance type includes: 1) HSA-HDHP without PDL; 2), HSA-HDHP with PDL; and 3) traditional plan.

Other co-variates include baseline asthma severity, co-morbidity, presence of other chronic conditions, self-reported and geocoded race/ethnicity data, neighborhood education and poverty levels, sex, age, state, individual versus family plan, baseline number of outpatient visits, presence of an inpatient hospitalization, total expenditures, employer size, average employer baseline expenditures per capita, number of family members, mean age of children in the family, mean age of adults, baseline mean family morbidity score, number of family members with asthma, number of asthma and other medications used by the family, and number of family ED visits and hospitalizations in the baseline year.

Analysis plan

Aim 1

The study team will analyze qualitative data in iterative cycles of content analysis in the manner described by Patton. In the second, deductive phase of analysis, investigators will consider data code-by-code to identify areas of convergence and divergence by insurance type.

Aim 2

Analyses will compare changes in outcomes from baseline to up to three years of follow-up among 1) asthma patients switched to HSA-HDHPs without PDLs from traditional plans vs. matched patients whose employers remain in traditional plans; and 2) patients switched to HSA-HDHPs with PDLs from HSA-HDHPs without PDLs vs. matched controls remaining in HSA-HDHPs without PDLs. The investigators will use separate regression models to compare year-to-year changes for each intervention group relative to its matched control group, rather than including all patients in a single model with multiple interaction terms.

The analyses will use both Interrupted Time Series (ITS) and Difference-in-Differences (DiD) frameworks. Controlling for potential confounders, analyses will use generalized linear models (GLMs) to model the independent effect of switching to each of the two types of HSA-HDHPs (with or without PDLs) on the likelihood of each outcome, assessed by interacting insurance type and study period variables in models. Extended GLMs - generalized estimating equations (GEE) and generalized linear mixed models (GLMM) - are appropriate methods to adjust for correlation within families and to examine changes in outcomes between baseline and follow-up.

This study will examine controller medication adherence using ITS. Investigators will test the statistical significance of level or trend changes following insurance plan type switch using GLM models, adjusting for seasonality and first-order autocorrelation between sequential monthly measurements using the empirical sandwich estimator.

For analyses of rescue medication use, investigators will focus on albuterol and levalbuterol inhaler users. The standardized number of rescue inhalers dispensed will be modeled as count data in difference-in-differences models. ITS models will be used to model changes in level and trend of monthly rates of rescue inhalers dispensed, as in previous studies. Analyses will also model the ratio of controller medications to total asthma medications. For analyses of asthma-related ED visits and hospitalizations, outcomes can be binary, counts, or continuous. The investigators will use logistic GEE models to estimate the effect of switching to each type of HSA-HDHP on binary outcomes such as any asthma-related hospitalization. Negative binomial regression will be used to model the effect for count outcomes such as ED visits. Investigators will select the conditional mean and variance functions based on the actual data, using a log link with a Gamma error distribution.

To determine the impact of HSA-HDHP with and without PDLs on vulnerable populations and test for heterogeneity of treatment effects among vulnerable populations, the investigators will first perform stratified analyses, comparing outcomes between intervention and control subgroups defined by the binary measures of the risk factors of interest (low income, minority race/ethnicity, moderate-severe asthma, presence of other chronic conditions, high morbidity based on the Johns Hopkins Adjusted Clinical Groups (ACG) system). Analyses will use three-way interaction terms (insurance type * study period * subgroup) to test for statistical differences between subgroups in the impact of the change to an HSA-HDHP with PDL vs. remaining in a traditional plan. In Aim 2 analyses, the investigators will include both adults and children together, with age included as a co-variate.

Aim 3

Analyses will use the same population, outcomes, study group comparisons, and modeling strategies as Aims 1 and 2 except that stratified analyses will be performed, comparing outcomes between intervention and control groups stratified by adult/child status. To statistically test for heterogeneity of treatment effect for adults vs. children, analyses will use three-way interaction terms (insurance type * study period * adult/child) to test for statistical differences between adults and children in the impact of the change to an HSA-HDHP with PDL vs. remaining in a HSA-HDHP without PDL. Analyses will be done at the individual level, but will include family-level variables as predictors of interest. Separately for adults and children, the investigators will test the extent to which having another family member with asthma, another chronic condition, or high baseline family ACG morbidity modifies the impact of HDHPs and PDLs on study outcomes for an individual asthma patient. The primary predictor of interest will be the interaction between the family-level variable, study period, and study group.

Aim 4

Analyses will be similar to those of Aim 2, but for OOP cost outcomes. The primary analyses of changes in OOP costs will use a DiD analytic framework. The investigators will follow the same approaches as used in analyzing ED visits and hospitalizations, employing two-part models/zero-inflated negative binomial models to account for zero costs. GEE or GLMM models will be used to examine changes in outcomes between baseline and follow-up to model the independent effect of switching to each of the two types of HSA-HDHPs (with or without PDLs) on the likelihood of having financial burden (OOP cost greater than 5% of income).

ELIGIBILITY:
Inclusion Criteria:

* adult or child with asthma, defined as having one outpatient claim, one emergency department claim, or one inpatient claim with an ICD-9/10 diagnosis code for asthma in the baseline period
* has employer-sponsored insurance from an employer who offers only one plan
* at least 24 months of continuous enrollment with pharmacy benefits between 2004 - 2017

Exclusion Criteria:

* other co-morbid pulmonary conditions identified in claims data (cystic fibrosis, immunodeficiency, bronchiectasis, congestive heart failure, pulmonary hypertension, or pulmonary embolism)
* enrolled through an employer who offers a choice of health insurance plans

Ages: 4 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Adults and children with asthma enrolled in an employer-sponsored plan from a large national insurance carrier between 2004 - 2017.
Sampling Method: Non-Probability Sample
Enrollment: 12238 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alison A Galbraith, MD, MPH, Principal Investigator — Harvard Pilgrim Health Care Institute
Locations (1):
- Harvard Pilgrim Health Care, Wellesley, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Note that Aim 1 of the project was a qualitative study with a separate protocol under the larger project approved by the IRB, and recruited entirely separate participants from the other Aims.
Pre-assignment Details: Aims 2 was an observational cohort study using pre-existing secondary claims data, not a clinical trial. After the study began, we found that we lacked a large enough sample of enrollees in the existing database who were eligible for the "traditional plan" arm. After approval from the funder, we modified the protocol to include a "HDHP without PDL" arm instead; thus the "traditional plan" group was not considered enrolled and we did not collect outcome data for this group.
Groups:
- HDHP With PDL: Enrollees switched from a high-deductible health plan (HDHP) without a preventive drug list (PDL) to a HDHP with a PDL
  HDHP with PDL: Enrollment in a Health Savings Account-eligible high-deductible health plan with an annual individual deductible of >$1000 that includes a preventive drug list (a list of certain chronic medications that are exempt from the deductible)
- HDHP Without PDL: Enrollees stayed in a high-deductible health plan (HDHP) without a preventive drug list (PDL).
Period: Overall Study
Arm/Group | HDHP With PDL | HDHP Without PDL
Started | 6087 | 6151
Completed | 6087 | 6151
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: HDHP with PDL group and matched control group (HDHP without PDL), unweighted. Note: after the study began, we found that we lacked a large enough sample size of enrollees eligible for the "traditional plan" arm. After discussion and approval from the funder, we changed to using a differently defined study arm with a larger sample size (the "HDHP without PDL" arm).
Groups:
- HDHP With PDL: Enrollees switched from a high-deductible health plan (HDHP) to a HDHP with a preventive drug list (PDL)
  HDHP with PDL: Enrollment in a Health Savings Account-eligible high-deductible health plan with an annual individual deductible of >$1000 that includes a preventive drug list (a list of certain chronic medications that are exempt from the deductible)
- HDHP Without PDL: Enrollees who stayed in a HDHP without a PDL.
- Total: Total of all reporting groups
Arm/Group | HDHP With PDL | HDHP Without PDL | Total
Number analyzed (Participants) | 6087 | 6151 | 12238
Age, Customized [Count of Participants; unit: Participants]
  Age (years): 4-17 | 987 | 976 | 1963
  Age (years): 18-29 | 1289 | 1313 | 2602
  Age (years): 30-39 | 729 | 952 | 1681
  Age (years): 40-49 | 1174 | 1231 | 2405
  Age (years): 50-64 | 1908 | 1679 | 3587
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3377 | 3447 | 6824
  Male | 2710 | 2704 | 5414
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/ethnicity: Asian, Non-Hispanic | 137 | 157 | 294
  Race/ethnicity: Black, Non-Hispanic | 365 | 361 | 726
  Race/ethnicity: Hispanic | 422 | 343 | 765
  Race/ethnicity: Other/unknown | 290 | 255 | 545
  Race/ethnicity: Non-Hispanic White | 4873 | 5035 | 9908
Any controller medication fill during baseline [Count of Participants; unit: Participants]
  Any controller fill | 1098 | 1146 | 2244
  No controller fill | 4989 | 5005 | 9994

OUTCOME MEASURES:

1. Primary Outcome: Change in Percentage of Days Covered for Inhaled Corticosteroids
Description: Adjusted mean change in adherence for inhaled corticosteroid medications as measured by change in percentage of days covered (PDC), relative to change in PDC for controls
Time Frame: baseline year to follow up year
Population: Participants with any fill in the baseline period. In this difference-in-differences study design, the outcome was the difference between arms in the difference in mean PDC from baseline to follow up. Note: after the study began, we found inadequate sample size for the "traditional plan" arm. After approval from the funder, we changed to using a differently defined study arm with a larger sample size (the "HDHP without PDL" arm) and did not collect outcome data for the "traditional plan" group.
Measure: Mean (95% Confidence Interval); unit: percentage of days
Arm/Group | HDHP With PDL | HDHP Without PDL
Number analyzed (Participants) | 135 | 140
percentage of days
  baseline period | 51.5 [47.0 to 56.1] | 44.7 [36.4 to 52.9]
  follow up period | 37.0 [31.6 to 42.5] | 29.1 [21.3 to 36.9]
Statistical Analysis 1: Comparison: HDHP With PDL vs HDHP Without PDL; Test type: Superiority; p = 0.05, GEE models; Negative binomial regression with GEE model; term of interest was interaction between study group and time period (baseline vs follow-up year); Mean Difference (Net) = 3.4, 95% CI 2-sided [-5.2 to 12.1] — Using terms from the regression model, we applied marginal effects methods to calculate mean adjusted baseline and follow-up PDC and absolute changes

2. Primary Outcome: Change in Percentage of Days Covered for Leukotriene Inhibitors
Description: Adjusted mean change in adherence for leukotriene inhibitor medications as measured by change in percentage of days covered (PDC), relative to change in PDC for controls
Time Frame: baseline year to follow up year
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: percentage of days
Arm/Group | HDHP With PDL | HDHP Without PDL
Number analyzed (Participants) | 389 | 392
percentage of days
  baseline period | 70.3 [67.8 to 72.8] | 72.7 [68.0 to 77.4]
  follow up period | 58.4 [54.9 to 62.0] | 59.1 [52.6 to 65.6]
Statistical Analysis 1: Comparison: HDHP With PDL vs HDHP Without PDL; Test type: Superiority; p = 0.05, GEE model; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 1.3, 95% CI 2-sided [-4.4 to 7.0] — [estimate comment as in outcome 1, analysis 1]

3. Primary Outcome: Change From Baseline in Percentage of Days Covered for Inhaled Corticosteroid-long-acting Beta Agonist Medications
Description: Adjusted mean change in adherence for Inhaled Corticosteroid-Long-Acting Beta Agonist medications as measured by change in percentage of days covered (PDC), relative to change in PDC for controls
Time Frame: baseline year to follow up year
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: percentage of days
Arm/Group | HDHP With PDL | HDHP Without PDL
Number analyzed (Participants) | 234 | 237
percentage of days
  baseline period | 55.9 [52.8 to 59.0] | 58.6 [54.3 to 62.8]
  follow up period | 44.3 [40.3 to 48.2] | 40.1 [33.8 to 46.4]
Statistical Analysis 1: Comparison: HDHP With PDL vs HDHP Without PDL; Test type: Superiority; p = 0.05, GEE model; Binomial regression with GEE model; term of interest was interaction between study group and time period (baseline vs follow-up year); Mean Difference (Net) = 6.0, 95% CI 2-sided [0.7 to 11.3] — [estimate comment as in outcome 1, analysis 1]

4. Primary Outcome: Asthma-related Emergency Department (ED) Visits
Description: Absolute change in asthma-related ED visits per 100 patients relative to controls
Time Frame: baseline year to follow up year
Population: Participants with persistent asthma in the baseline period. In this difference-in-differences design, the outcome was the difference between arms in the difference in mean rates of ED visits from baseline to follow up. Note: after the study began, we found inadequate sample size for the "traditional plan" arm. After approval from the funder, we changed to using a study arm with a larger sample size (the "HDHP without PDL" arm) and did not collect outcome data for the "traditional plan" group.
Measure: Mean (95% Confidence Interval); unit: ED visits per 100 patients
Arm/Group | HDHP With PDL | HDHP Without PDL
Number analyzed (Participants) | 6087 | 6087
ED visits per 100 patients
  baseline period | 2.29 [1.90 to 2.68] | 2.48 [1.72 to 3.25]
  follow up period | 2.10 [1.72 to 2.47] | 2.10 [1.56 to 2.65]
Statistical Analysis 1: Comparison: HDHP With PDL vs HDHP Without PDL; Test type: Superiority; p = 0.05, GEE model; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 0.16, 95% CI 2-sided [-0.74 to 1.06] — [estimate comment as in outcome 1, analysis 1]

5. Primary Outcome: Out-of-pocket Costs
Description: change in out-of-pocket (OOP) costs for asthma medications and other health services
Time Frame: baseline year to follow up year
Population: Patients with persistent asthma in the baseline period. In this difference-in-differences study design, the outcome was the difference between arms in the difference in mean OOP costs from baseline to follow up. Note: after the study began, we found inadequate sample size for the "traditional plan" arm. After approval from the funder, we changed to using a study arm with a larger sample size (the "HDHP without PDL" arm) and did not collect outcome data for the "traditional plan" group.
Measure: Mean (95% Confidence Interval); unit: dollars
Arm/Group | HDHP With PDL | HDHP Without PDL
Number analyzed (Participants) | 6087 | 6087
dollars
  baseline period | 130 [121 to 138] | 122 [110 to 133]
  follow up period | 85 [79 to 92] | 112 [100 to 124]
Statistical Analysis 1: Comparison: HDHP With PDL vs HDHP Without PDL; Test type: Superiority; p = 0.05, GEE model; [statistical method as in outcome 1, analysis 1]; Median Difference (Net) = -34, 95% CI 2-sided [-47 to -21] — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: Adverse events information was not collected.
Description: Adverse events information was not collected.
Groups:
- HDHP Without PDL: Enrollees switched from a traditional plan to a high-deductible health plan (HDHP) without a preventive drug list (PDL). Enrollees who stayed in a HDHP without a PDL will also serve as controls for the study group who switch from HDHPs without PDLs to HDHPs with PDLs.
Arm/Group | HDHP With PDL | HDHP Without PDL
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-16): https://cdn.clinicaltrials.gov/large-docs/36/NCT03175536/Prot_SAP_000.pdf